CLINICAL TRIAL: NCT02920385
Title: A Trial Investigating the Influence of Oral Semaglutide on the Pharmacokinetics of Levothyroxine and the Influence of Co-administered Tablets on the Pharmacokinetics of Semaglutide Administered Orally in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4279; 2015-005558-36 (EudraCT Number); U1111-1177-2807 (Other: WHO)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levothyroxine/SNAC/Placebo/Semaglutide (Experimental)
  Interventions: Drug: Semaglutide; Drug: SNAC; Drug: Levothyroxine; Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Oral administration once daily alone or together with levothyroxine or Placebo
Drug: SNAC — Oral administration once daily alone or together with levothyroxine or semaglutide
Drug: Levothyroxine — Oral administration alone or together with SNAC or oral semaglutide
Drug: Placebo — Oral administration once daily together with semaglutide

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the influence of oral semaglutide on the pharmacokinetics (the exposure of the trial drug in the body) of levothyroxine and the influence of co-administered tablets on the pharmacokinetics of semaglutide administered orally in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-50 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) 20.0 to 29.9 kg/m^2 (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Smoker (defined as a subject who is smoking at least 1 cigarette or the equivalent per day)
* Unable or unwilling to refrain from smoking and use of nicotine substitute products within 48 hours prior to and during the inpatient periods
* Any blood draw in excess of 25 mL in the past 30 days, or donation of blood or plasma in excess of 400 mL within the 90 days preceding screening
* History (as declared by the subject) of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* History (as declared by the subject) or presence of clinical or non-clinical thyroid disease, including thyroid palpation abnormalities, levels of T3 or T4 (total and free) or TSH outside reference limits, or presence of thyroid antibodies (Thyroid Stimulating Hormone Receptor Antibody, Thyroperoxidase Antibody or Thyroid Antithyroglobulin Antibodies)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Baseline-corrected area under the total T4 serum concentration-time curve from 0 to 48 hours after a single dose of levothyroxine | On day 1 (levothyroxine administered alone), on day 38 (levothyroxine co-administered with SNAC) and on day 89 (levothyroxine co-administered with oral semaglutide)
Area under the semaglutide plasma concentration-time curve during a dosing interval (0-24 hours) at steady state | On day 88 (oral semaglutide administered alone) and on day 139 (oral semaglutide co-administered with placebo tablets)

SECONDARY OUTCOMES:
Baseline-corrected maximum observed total T4 serum concentration from 0 to 48 hours after a single dose of levothyroxine | On day 1 (levothyroxine administered alone), on day 38 (levothyroxine co-administered with SNAC) and on day 89 (levothyroxine co-administered with oral semaglutide)
Maximum observed semaglutide plasma concentration during a dosing interval from (0-24 hours) at steady state | On day 88 (oral semaglutide administered alone) and on day 139 (oral semaglutide co-administered with placebo tablets)
Area under the SNAC plasma concentration-time curve during a dosing interval (0-24 hours) at steady state | On day 88 (oral semaglutide administered alone) and on day 139 (oral semaglutide co-administered with placebo tablets)
Maximum observed SNAC plasma concentration during a dosing interval (0-24 hours) at steady state | On day 88 (oral semaglutide administered alone) and on day 139 (oral semaglutide co-administered with placebo tablets)

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to Novo Nordisk disclosure commitment on novonordisk-trials.com